CLINICAL TRIAL: NCT02850289
Title: A Prospective Study of Peginterferon Alfa-2a and Ribavirin: Outcomes Assessment in Chronic Hepatitis C Patients
Brief Title: APPROACH Study: Quality of Life and Outcomes Assessment in Participants With Chronic Hepatitis C (CHC) Treated With Pegylated Interferon (PEG-IFN) Alfa-2a and Ribavirin
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20090
Record Dates: First submitted 2016-07-28; First posted 2016-07-29 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pegylated Interferon (PEG-IFN) alfa-2a and Ribavirin: Participants with hepatitis C who were to be treated with combination of pegylated interferon (PEG-IFN) alfa-2a and ribavirin, within 7 days of baseline, with ongoing management at investigator's discretion.
  Interventions: Drug: Pegylated interferon (PEG-INF) alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon (PEG-INF) alfa-2a — Pegylated interferon (PEG-IFN) alfa-2a will be administered as per investigator's discretion and will be in line with the current product monograph.
  Other Names: PEGASYS
Drug: Ribavirin — Ribavirin will be administered as per investigator's discretion and will be in line with the current product monograph.
  Other Names: COPEGUS

SUMMARY:
This multi-center, observational study will examine the clinical use and outcomes of pegylated interferon (PEG-IFN) alfa-2a and ribavirin combination (PEGASYS RBV) in participants with chronic hepatitis C (CHC). Study visits will be scheduled for baseline, 12, 24 and 48 weeks after baseline. An additional follow-up visit at week 72 will be required for participants with an HCV genotype other than 2 or 3. Quality of life data will be collected at baseline, and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for and scheduled to receive treatment with commercially available PEG-IFN alfa-2a and ribavirin combination
* Serologic evidence of chronic hepatitis C (CHC) infection
* Detectable serum hepatitis C virus - ribonucleic acid (HCV-RNA)
* Negative urine or blood pregnancy test
* Fertile participants receiving treatment to use two forms of effective contraception during treatment and for 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or who are breast feeding, or male partners of women who are pregnant
* Received any investigational drug less than or equal to (</=) 6 weeks prior to enrollment
* Moderate hepatic failure [Child-Pugh greater than or equal to (>/=) B]
* Co-infection with human immunodeficiency virus (HIV) or hepatitis B
* Autoimmune hepatitis
* Known hypersensitivity to alfa interferons, E. coli-derived products, polyethylene glycol, ribavirin and/or any ingredient in the formulation or component of PEG-IFN alfa-2a or ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with hepatitis C, who were to be treated with combination of pegylated interferon (PEG-IFN) alfa-2a and ribavirin (PEGASYS RBV), within 7 days of baseline.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Sustained Virologic Response (SVR) | Up to Week 72

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36) Physical Composite Score | Baseline, Week 12, 24, 48 and 72
Short Form Health Survey (SF-36) Mental Composite Score | Baseline, Week 12, 24, 48 and 72
Percentage of Participants with Adverse Events of Special Interest Leading to Study Medication Discontinuation | Up to Week 72
Percentage of Participants Who Utilized Resources | Baseline, Week 12, 24, 48 and 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- Canada (28):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Vernon, British Columbia
  - West Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Barrie, Ontario
  - Brampton, Ontario
  - Downsview, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Richmond Hill, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan